CLINICAL TRIAL: NCT01066117
Title: Effectiveness of PeeRelease - a Gel Absorbent Pad in Moderate to Severe Urinary Incontinence Over Existing Solutions
Brief Title: Effectiveness of PeeRelease - a Gel Absorbent Pad in Moderate to Severe Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tisteron Ltd. (Industry)
Responsible Party: Tisteron Ltd, Tisteron Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5481
Record Dates: First submitted 2010-02-04; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinent
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: PeeRelease gel absorbent pad — A larger gel containing pad was developed, suitable to absorb up to half a liter liquid, it eliminates odors and enables the users to wear ordinary clothes

SUMMARY:
The purpose of the proposed study is to test the effect of the new gel pad on the quality of life of urinary incontinent men and women and to assess to what extent the gel pad improves the quality of life of incontinence persons.

DETAILED DESCRIPTION:
The devices available today on the market serve two polar incontinence conditions: those who have severe urinary incontinence and need to use diapers several times per day, or those who have mild urinary incontinence and can use pads.

Such circumstances call for a search of new solution that may provide the benefit of freeing those with moderate incontinence from changing pads several times a day or staying constantly very near a bathroom, as well as freeing those with severe incontinence from using cumbersome diapers.

A larger gel containing pad was developed, suitable to absorb up to half a litter liquid, it eliminates odors and enables the users to wear ordinary clothes . It was presented for clinical trial.

The objectives of the clinical trial, proposed hereafter is to assess to what extent the new gel pad presents an advantage over the existing means of coping with urinary incontinence in cases when medicinal treatment or surgery is not appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Urinary incontinent women and men who loose urine at a quantity higher than drops (50CC or more).
2. Three segments of such persons will be included in the study:

   * pregnant women who are temporary urinary incontinent
   * women of the age 40+ who are urinary incontinent
   * men who are urinary incontinent (post prostatectomy)

Exclusion Criteria:

1. Urinary incontinent disabled patients who need nursing
2. Patients who presently have cancer of any kind,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Significant improvement in quality of life for men and women who use the new gel pad in comparison to usage of existing solutions; this means a difference of at least 5 scores on the 1-100 I-QoL score scale | two weeks

SECONDARY OUTCOMES:
Pad weight and number of pads used per day | daily
Observation for any development of rash due to patients' sensitivity to the pad | two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel